CLINICAL TRIAL: NCT05190419
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2b Dose-Ranging Study to Evaluate the Efficacy and Safety of Orismilast in Adults With Moderate-to-Severe Plaque-Type Psoriasis
Brief Title: Study to Assess the Efficacy and Safety of Orismilast in Psoriasis
Acronym: IASOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNI50001-203; 2021-003209-22 (EudraCT Number)
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis; Skin Diseases
Keywords: Psoriasis; Orismilast
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly in a 1:1:1:1 ratio to receive 1 of the 3 orismilast modified release doses (20 mg, 30 mg, or 40 mg) or placebo twice daily (BID)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Tablets will be packaged in the same type of blister and the active and placebo tablets will have the same appearance (in terms of size, form, weight, and color).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orismilast modified release tablets 20 mg BID (Experimental): Oral, twice daily morning and evening for 16 weeks
  Interventions: Drug: Orismilast modified release tablets
- Orismilast modified release tablets 30 mg BID (Experimental): Oral, twice daily morning and evening for 16 weeks
  Interventions: Drug: Orismilast modified release tablets
- Orismilast modified release tablets 40 mg BID (Experimental): Oral, twice daily morning and evening for 16 weeks
  Interventions: Drug: Orismilast modified release tablets
- Placebo tablets BID (Placebo Comparator): Oral, twice daily morning and evening for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orismilast modified release tablets — Orismilast modified release is a next generation phosphodiesterase-4 (PDE4) inhibitor with high selectivity for the PDE4 subtypes linked to inflammation.
  Other Names: UNI50001; LEO32731
  Arms: Orismilast modified release tablets 20 mg BID; Orismilast modified release tablets 30 mg BID; Orismilast modified release tablets 40 mg BID
Drug: Placebo — Matching placebo tablets
  Arms: Placebo tablets BID

SUMMARY:
This study investigates 3 different doses of orismilast modified release compared to placebo in adult patients with moderate-to-severe plaque-type psoriasis. The purpose of the study is to assess the effect of orismilast modified release in moderate-to-severe plaque-type psoriasis and assess the safety aspects of these 3 different doses.The patients will receive an oral treatment of either orismilast modified release tablets or placebo tablets 2 times a day for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Male and female patients ≥18 years of age
3. Body weight of >40 kg
4. Diagnosis of chronic, stable plaque-type psoriasis. If the patient is diagnosed with psoriasis arthritis, the arthritis should be stable.
5. Moderate-to-severe plaque-type psoriasis as defined by Psoriasis Activity and Severity Index (PASI) ≥12, body surface area (BSA) ≥10%, and Investigator Global Assessment (IGA) ≥3.
6. Candidate for systemic antipsoriatic treatment or phototherapy.

Exclusion Criteria:

1. Therapy-resistant psoriasis
2. Unstable psoriasis or psoriatic arthritis with acute deterioration within 4 weeks of the Screening visit.
3. History of allergy or hypersensitivity to any component of the study treatment.
4. Active infection (eg, bacteria, viral, fungal) requiring treatment with systemic antibiotics within 4 weeks of the Screening visit.
5. Malignancy or history of malignancy except for treated (ie, cured) basal cell skin carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. A., MD, Study Director — UNION therapeutics A/S
Locations (34):
- United States (7):
  - Central Connecticut Dermatology, Cromwell, Connecticut
  - GWU MFA, Washington D.C., District of Columbia
  - ALLCUTIS Research, LLC, Beverly, Massachusetts
  - ALLCUTIS Research, LLC, Portsmouth, New Hampshire
  - Bruce E. Katz, MD, New York, New York
  - Sadick Research Group LLC, New York, New York
  - Apex Clinical Research Center, Mayfield Heights, Ohio
- Germany (12):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Rosenpark Research GmbH, Darmstadt
  - Hautarztpraxis Dr.Gerlach, Dresden
  - Derma-Study-Center-Friedrichshafen, Friedrichshafen
  - Klinische Forschung Hamburg GmbH, Hamburg
  - TFS Trial From Support GmbH, Hamburg
  - MVZ DermaKiel GmbH, Kiel
  - Studienzentrum Dr.Beate Schwarz, Langenau
  - Hautarztpraxis Mahlow, Mahlow
  - LMU Muenchen, Klinik und Poliklinik fur Dermatologie und Allergologie, München
  - KliFOs - Klinische Forschung Osnabrueck, Osnabrück
- Poland (14):
  - NZOZ Specjalistyczny Orodek Dermatologiczny DERMAL, Bialystok
  - Specjalistyczna Praktyka Lekarska Gabinet Dermatologiczny dr n.med. Edyta Gebska, Chorzów
  - Zespol Naukowo - Leczniczy Dermatologiczne Centrum Uzdrowiskowe Iwolang Sp. z o.o., Iwonicz-Zdrój
  - Provita Sp. z o.o., Katowice
  - Centrum Medyczne All-Med, Krakow
  - Klinika Badawcza, Malbork
  - Laser Clinic, Szczecin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o. o., Tarnów
  - High-Med.Przychodnia Specjalistyczna, Warsaw
  - Klinika Ambroziak, Warsaw
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
  - dermMedica Sp z.o.o, Wroclaw
  - Wromedica, Wroclaw
- Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warren RB, Weiss A, Felding J, Sommer MOA, Garcet S, Krueger JG. Orismilast, a Potent and Selective PDE4B/D Inhibitor, Reduces Protein Levels of Key Disease Driving Cytokines in the Skin of Patients With Plaque Psoriasis. Exp Dermatol. 2025 Sep;34(9):e70153. doi: 10.1111/exd.70153. PMID 40970551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 202 participants were randomized at 26 sites in Germany (8 sites), Poland (12 sites), the United Kingdom (1 site), and the US (5 sites).
Groups:
- Orismilast Modified Release Tablets 30 mg BID; Orismilast Modified Release Tablets 40 mg BID: Oral, twice daily morning and evening for 16 weeks
  Orismilast modified release tablets: Orismilast modified release is a next generation PDE4 inhibitor with high selectivity for the PDE4 subtypes linked to inflammation.
Period: Overall Study
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Started | 51 | 48 | 50 | 53
Completed | 32 | 34 | 33 | 26
Not Completed | 19 | 14 | 17 | 27
Not completed — Lack of Efficacy | 8 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 1 | 2 | 2
Not completed — Adverse Event | 2 | 10 | 11 | 21
Not completed — Lost to Follow-up | 1 | 2 | 3 | 1
Not completed — Other | 1 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Groups:
- Orismilast Modified Release Tablets 20 mg BID; Orismilast Modified Release Tablets 30 mg BID; Orismilast Modified Release Tablets 40 mg BID: Oral, twice daily morning and evening for 16 weeks
  Orismilast modified release tablets: Orismilast modified release is a next generation PDE4 inhibitor with high selectivity for the PDE4 subtypes linked to inflammation.
- Total: Total of all reporting groups
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID | Total
Number analyzed (Participants) | 51 | 48 | 50 | 53 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.10 (11.98) | 45.40 (13.87) | 48.20 (13.40) | 44.30 (14.60) | 45.70 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 11 | 15 | 55
  Male | 39 | 31 | 39 | 38 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 1 | 5
  Not Hispanic or Latino | 49 | 48 | 48 | 52 | 197
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 43 | 46 | 47 | 180
  Black or African American | 0 | 0 | 0 | 1 | 1
  Other | 2 | 0 | 0 | 0 | 2
  Not reported | 5 | 5 | 4 | 5 | 19
Psoriatic Arthritis [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 5 | 6 | 14
  No | 50 | 46 | 45 | 47 | 188
Disease duration [Mean (Standard Deviation); unit: years] | 19.30 (11.33) | 22.00 (14.21) | 18.10 (11.99) | 19.80 (13.69) | 19.80 (12.83)
Disease duration > 2 years [Count of Participants; unit: Participants]
  Yes | 49 | 47 | 47 | 49 | 192
  No | 2 | 1 | 3 | 4 | 10
Height [Mean (Standard Deviation); unit: cm] | 176.26 (8.67) | 174.14 (8.78) | 173.87 (9.30) | 176.90 (8.57) | 175.33 (8.86)
Weight [Mean (Standard Deviation); unit: kg] | 91.48 (20.33) | 94.85 (29.96) | 91.65 (16.17) | 91.08 (21.17) | 92.22 (22.24)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.420 (6.271) | 31.019 (8.548) | 30.464 (5.963) | 29.000 (5.921) | 29.948 (6.727)
Females of Child-bearing potential [Count of Participants; unit: Participants] — Population: Number of participants analyzed includes the total number of females of child-bearing potential in each arm.
  Participants
    Yes: number analyzed (Participants) | 12 | 17 | 11 | 15 | 55
    Yes | 10 | 13 | 5 | 10 | 38
    No: number analyzed (Participants) | 12 | 17 | 11 | 15 | 55
    No | 2 | 4 | 6 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Psoriasis Activity and Severity Index (PASI) Score at Week 16
Description: The Psoriasis Activity and Severity Index (PASI) is a measure of psoriatic disease severity, taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI.
Time Frame: Baseline and Week 16
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percent change | -17.30 (7.07) | -52.60 (6.80) | -61.20 (6.67) | -63.70 (6.96)
Statistical Analysis 1: Comparison: Placebo Tablets BID vs Orismilast Modified Release Tablets 20 mg BID; Test type: Superiority; p < 0.001, ANCOVA — No adjustment for multiplicity was made and the 0.05 level of significance was used to claim efficacy compared with placebo; p-value is calculated by analysis of covariance with treatment group as factor and baseline PASI as covariate; Mean Difference (Net) = -35.4, 95% CI 2-sided [-54.7 to -16.0], Standard Error of Mean 9.83
Statistical Analysis 2: Comparison: Placebo Tablets BID vs Orismilast Modified Release Tablets 30 mg BID; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; p-value is calculated by analysis of covariance with treatment group as factor and baseline PASI as covariate; Mean Difference (Net) = -43.9, 95% CI 2-sided [-63.1 to -24.8], Standard Error of Mean 9.75
Statistical Analysis 3: Comparison: Placebo Tablets BID vs Orismilast Modified Release Tablets 40 mg BID; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; p-value is calculated by analysis of covariance with treatment group as factor and baseline PASI as covariate; Mean Difference (Net) = -46.4, 95% CI 2-sided [-65.6 to -27.3], Standard Error of Mean 9.75

2. Secondary Outcome: Percentage of Participants Who Achieved 75% Reduction in PASI (PASI75) Response at Week 16
Description: The PASI is a measure of psoriatic disease severity, taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI. PASI75 is 75% reduction from Baseline in PASI score.
Time Frame: At Week 16
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percentage of participants
  Yes | 16.5 | 39.5 | 49.0 | 46.4
  No | 83.5 | 60.5 | 51.0 | 53.6

3. Secondary Outcome: Percentage of Participants Who Achieved a Score of Clear (0) or Almost Clear (1) and an at Least 2-point Improvement in Investigator Global Assessment (IGA) at Week 16
Description: The IGA is a measure used by physicians to determine the patient's overall severity of disease. The static version is used in this trial for measurement at a single point in time as indicated in the schedule of assessments. The investigator will rate the severity of patient's psoriasis on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: At Week 16
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percentage of participants
  Yes | 6.9 | 26.2 | 24.5 | 20.6
  No | 93.1 | 73.8 | 75.5 | 79.4

4. Secondary Outcome: Percentage of Participants Who Achieved a Score of Clear (0) or Almost Clear (1) and an at Least 2-point Improvement in Investigator Global Assessment (IGA) at Weeks 4, 8, 12, and 20
Description: as for outcome 3
Time Frame: At Weeks 4, 8, 12, and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percentage of participants
  Week 4, Yes | 2.1 | 4.2 | 4.3 | 4.1
  Week 4, No | 97.9 | 95.8 | 95.7 | 95.9
  Week 8, Yes | 0 | 10.9 | 17.0 | 8.4
  Week 8, No | 100 | 89.1 | 83.0 | 91.6
  Week 12, Yes | 4.6 | 25.4 | 23.4 | 17.6
  Week 12, No | 95.4 | 74.6 | 76.6 | 82.4
  Week 20, Yes | 11.3 | 21.0 | 11.1 | 10.8
  Week 20, No | 88.7 | 79.0 | 88.9 | 89.2

5. Secondary Outcome: Percentage of Participants Who Achieved 75% Reduction in PASI (PASI75) Response at Weeks 4, 8, 12, and 20
Description: as for outcome 2
Time Frame: At Weeks 4, 8, 12, and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percentage of participants
  Week 4, Yes | 6.0 | 8.4 | 10.8 | 9.6
  Week 4, No | 94.0 | 91.6 | 89.2 | 90.4
  Week 8, Yes | 11.8 | 32.5 | 37.0 | 31.2
  Week 8, No | 88.2 | 67.5 | 63.0 | 68.8
  Week 12, Yes | 12.3 | 42.5 | 49.5 | 38.5
  Week 12, No | 87.7 | 57.5 | 50.5 | 61.5
  Week 20, Yes | 18.7 | 31.6 | 22.0 | 29.7
  Week 20, No | 81.3 | 68.4 | 78.0 | 70.3

6. Secondary Outcome: Percentage of Participants Who Achieved 50%, 90%, and 100% Reduction in PASI Response at Weeks 4, 8, 12, 16, and 20
Description: The PASI is a measure of psoriatic disease severity, taking into account qualitative lesion characteristics (erythema, induration, and desquamation) and percentage of affected skin surface area on defined anatomical regions. PASI score ranges from 0 to 72, with higher scores reflecting greater disease severity. Erythema, induration/thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. The scores for each anatomic region are combined to yield the final PASI. PASI 50, 90, and 100 is 50%, 90%, and 100% reduction from Baseline in PASI score, respectively.
Time Frame: At Weeks 4, 8, 12, 16, and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
Participants
  Week 4, PASI 50 | 8 | 16 | 18 | 21
  Week 4, PASI 90 | 0 | 1 | 2 | 3
  Week 4, PASI 100 | 0 | 0 | 0 | 0
  Week 8, PASI 50 | 11 | 28 | 28 | 27
  Week 8, PASI 90 | 1 | 4 | 6 | 5
  Week 8, PASI 100 | 0 | 0 | 3 | 1
  Week 12, PASI 50 | 15 | 27 | 32 | 22
  Week 12, PASI 90 | 3 | 10 | 9 | 8
  Week 12, PASI 100 | 0 | 5 | 4 | 0
  Week 16, PASI 50 | 13 | 23 | 30 | 25
  Week 16, PASI 90 | 4 | 11 | 10 | 12
  Week 16, PASI 100 | 1 | 4 | 4 | 1
  Week 20, PASI 50 | 12 | 19 | 19 | 17
  Week 20, PASI 90 | 3 | 9 | 6 | 4
  Week 20, PASI 100 | 2 | 2 | 1 | 1

7. Secondary Outcome: Percent Change From Baseline in Psoriasis Activity and Severity Index (PASI) Score at Weeks 4, 8, 12, and 20
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, 12, and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
percent change
  Week 4 | -14.40 (4.33) | -35.40 (4.40) | -38.40 (4.43) | -38.70 (4.24)
  Week 8 | -16.10 (5.79) | -48.30 (5.76) | -54.20 (5.94) | -53.60 (5.87)
  Week 12 | -18.10 (6.61) | -56.10 (6.30) | -61.70 (6.40) | -57.50 (6.59)
  Week 20 | -13.70 (9.69) | -35.00 (9.11) | -30.50 (9.11) | -36.20 (10.57)

8. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Weeks 16 and 20
Description: The DLQI is a 10-item validated questionnaire completed by the patient used to assess the impact of skin disease on the patient's quality of life (QoL) during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0 to 3 ("not at all," "a little," "a lot," and "very much," respectively), giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL.
Time Frame: Baseline and Weeks 16 and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug. "n" represents the number of participants analyzed at each time point in each treatment arm.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 34 | 34 | 35 | 27
percent change
  Week 16 | -4.9 (1.02) | -8.8 (1.01) | -7.7 (1.00) | -7.3 (1.14)
  Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Week 20 | -5.1 (1.06) | -5.0 (1.02) | -4.0 (1.02) | -4.9 (1.17)

9. Secondary Outcome: Percent Change From Baseline in Affected Body Surface Area (BSA) at Weeks 4, 8, 12, 16, and 20
Description: The BSA assessment estimates the extent of disease or skin affected by psoriasis and is expressed as a percentage of total body surface. BSA was determined by the Investigator or designee using the patient palm = 1% BSA rule. The patient's palm is measured from the wrist to the proximal interphalangeal and thumb.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug. "n" represents the number of participants analyzed at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 46 | 50 | 52
percent change
  Week 4 | -2.30 (1.62) | -5.60 (1.69) | -7.20 (1.63) | -6.50 (1.59)
  Week 8: number analyzed (Participants) | 47 | 42 | 40 | 38
  Week 8 | -3.80 (1.67) | -9.20 (1.75) | -11.40 (1.77) | -11.60 (1.80)
  Week 12: number analyzed (Participants) | 38 | 38 | 36 | 29
  Week 12 | -5.30 (1.80) | -12.90 (1.81) | -14.70 (1.83) | -15.10 (2.00)
  Week 16: number analyzed (Participants) | 34 | 35 | 35 | 28
  Week 16 | -6.90 (1.87) | -13.50 (1.86) | -14.40 (1.85) | -18.10 (2.02)
  Week 20: number analyzed (Participants) | 30 | 34 | 33 | 26
  Week 20 | -6.20 (1.96) | -10.10 (1.88) | -8.10 (1.89) | -16.00 (2.08)

10. Secondary Outcome: Percent Change From Baseline in Total Score of Psoriasis Symptom Scale (PSS) at Weeks 4, 8, 12, 16, and 20
Description: The PSS is a 4-item patient-completed questionnaire (Rentz 2017). It is patient relevant, its domains are reliable and valid, and it takes few minutes to complete. The PSS assesses severity of pain, itching, redness, and burning during the past 24 hours using a 5-point severity scale from 0 = none to 4 = very severe.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 49 | 45 | 46 | 49
percent change
  Week 4 | -1.1 (3.82) | -4.6 (3.38) | -3.2 (3.77) | -3.8 (3.80)
  Week 8: number analyzed (Participants) | 46 | 41 | 39 | 37
  Week 8 | -1.8 (3.23) | -4.9 (3.61) | -5.2 (4.17) | -5.4 (3.91)
  Week 12: number analyzed (Participants) | 37 | 36 | 36 | 27
  Week 12 | -2.3 (3.46) | -6.2 (3.79) | -5.2 (4.28) | -5.5 (4.47)
  Week 16: number analyzed (Participants) | 34 | 35 | 35 | 27
  Week 16 | -1.8 (3.27) | -5.7 (4.25) | -4.8 (4.32) | -5.1 (3.48)
  Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Week 20 | -2.3 (3.20) | -2.9 (4.71) | -2.2 (4.84) | -3.1 (3.73)

11. Secondary Outcome: Percent Change From Baseline in Each Individual Item of Psoriasis Symptom Scale (PSS) at Weeks 4, 8, 12, 16, and 20
Description: as for outcome 10
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 20
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 50 | 45 | 49 | 50
percent change
  Pain, Week 4 | -0.6 (0.13) | -1.0 (0.14) | -0.5 (0.13) | -0.8 (0.13)
  Pain, Week 8: number analyzed (Participants) | 46 | 41 | 39 | 37
  Pain, Week 8 | -0.6 (0.14) | -0.9 (0.14) | -0.9 (0.14) | -1.0 (0.15)
  Pain, Week 12: number analyzed (Participants) | 37 | 36 | 36 | 27
  Pain, Week 12 | -0.6 (0.15) | -1.1 (0.15) | -0.9 (0.15) | -0.9 (0.17)
  Pain, Week 16: number analyzed (Participants) | 34 | 35 | 35 | 27
  Pain, Week 16 | -0.4 (0.15) | -1.0 (0.15) | -0.8 (0.15) | -0.7 (0.17)
  Pain, Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Pain, Week 20 | -0.5 (0.16) | -0.4 (0.15) | -0.2 (0.15) | -0.5 (0.17)
  Redness, Week 4 | -0.3 (0.13) | -1.0 (0.14) | -0.9 (0.13) | -0.9 (0.13)
  Redness, Week 8: number analyzed (Participants) | 46 | 41 | 39 | 37
  Redness, Week 8 | -0.6 (0.14) | -1.1 (0.14) | -1.3 (0.15) | -1.2 (0.15)
  Redness, Week 12: number analyzed (Participants) | 37 | 36 | 36 | 27
  Redness, Week 12 | -0.9 (0.15) | -1.5 (0.15) | -1.3 (0.15) | -1.2 (0.17)
  Redness, Week 16: number analyzed (Participants) | 34 | 35 | 35 | 27
  Redness, Week 16 | -0.6 (0.15) | -1.4 (0.15) | -1.2 (0.15) | -1.2 (0.17)
  Redness, Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Redness, Week 20 | -0.7 (0.16) | -0.7 (0.15) | -0.6 (0.15) | -0.9 (0.17)
  Itching, Week 4 | -0.4 (0.14) | -1.2 (0.14) | -0.8 (0.14) | -0.9 (0.14)
  Itching, Week 8: number analyzed (Participants) | 46 | 41 | 39 | 37
  Itching, Week 8 | -0.6 (0.14) | -1.3 (0.15) | -1.1 (0.15) | -1.2 (0.15)
  Itching, Week 12: number analyzed (Participants) | 37 | 36 | 36 | 27
  Itching, Week 12 | -0.5 (0.15) | -1.4 (0.16) | -1.2 (0.16) | -1.1 (0.17)
  Itching, Week 16: number analyzed (Participants) | 34 | 35 | 35 | 27
  Itching, Week 16 | -0.4 (0.16) | -1.3 (0.16) | -1.2 (0.16) | -0.9 (0.17)
  Itching, Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Itching, Week 20 | -0.7 (0.17) | -0.5 (0.16) | -0.5 (0.16) | -0.5 (0.18)
  Burning, Week 4 | -0.4 (0.14) | -1.2 (0.15) | -0.7 (0.14) | -0.7 (0.14)
  Burning, Week 8: number analyzed (Participants) | 46 | 41 | 39 | 37
  Burning, Week 8 | -0.7 (0.15) | -1.3 (0.15) | -1.0 (0.15) | -1.2 (0.16)
  Burning, Week 12: number analyzed (Participants) | 37 | 36 | 36 | 27
  Burning, Week 12 | -0.6 (0.16) | -1.4 (0.16) | -1.1 (0.16) | -1.1 (0.18)
  Burning, Week 16: number analyzed (Participants) | 34 | 35 | 35 | 27
  Burning, Week 16 | -0.5 (0.16) | -1.3 (0.16) | -1.1 (0.16) | -0.9 (0.18)
  Burning, Week 20: number analyzed (Participants) | 30 | 33 | 33 | 25
  Burning, Week 20 | -0.5 (0.17) | -0.5 (0.16) | -0.2 (0.16) | -0.4 (0.18)

12. Secondary Outcome: Percentage of Participants Who Experienced Psoriasis Rebound by Week 20
Description: as for outcome 1
Time Frame: At Week 20
Population: The intent-to-treat (ITT) population included all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
Number analyzed (Participants) | 51 | 48 | 50 | 53
Participants | 6 | 2 | 5 | 2

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo Tablets BID | Orismilast Modified Release Tablets 20 mg BID | Orismilast Modified Release Tablets 30 mg BID | Orismilast Modified Release Tablets 40 mg BID
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48 | 0/50 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/48 | 1/50 | 0/53
Other Adverse Events (participants affected / at risk) | 23/51 | 37/48 | 42/50 | 50/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablets BID (N=51) | Orismilast Modified Release Tablets 20 mg BID (N=48) | Orismilast Modified Release Tablets 30 mg BID (N=50) | Orismilast Modified Release Tablets 40 mg BID (N=53)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablets BID (N=51) | Orismilast Modified Release Tablets 20 mg BID (N=48) | Orismilast Modified Release Tablets 30 mg BID (N=50) | Orismilast Modified Release Tablets 40 mg BID (N=53)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 18 (24) | 24 (35) | 24 (43)
Nausea (Gastrointestinal disorders) | 2 (2) | 11 (12) | 19 (23) | 22 (24)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (9)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 6 (8)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (6) | 7 (19)
Headache (Nervous system disorders) | 3 (6) | 6 (9) | 13 (16) | 11 (14)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 7 (8) | 8 (10)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (3) | 1 (1) | 2 (2) | 3 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Slow response to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema migrans (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (2) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematocrit increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary sediment present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ultrasound abdomen abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT05190419/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT05190419/SAP_001.pdf